CLINICAL TRIAL: NCT02955446
Title: Compassionate Use Protocol for PF-03084014 in Patients With Advanced Solid Tumor Malignancies: Continuing Study Drug Administration in Desmoid Patients Receiving Clinical Benefit
Brief Title: Compassionate Use Protocol for PF-03084014 in Patients With Advanced Solid Tumor Malignancies
Status: No longer available | Type: Expanded Access
Sponsor: University of Colorado, Denver (Other)
Collaborators: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 15-2088.cc
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Neoplasm; Desmoid Tumor
Keywords: Refractory Tumors; Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms; Desmoid Tumors | interventions — nirogacestat

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: PF-03084014 — Two patients enrolled in this study will continue receiving 80mg BID doses of PF-03084014, which was the same dose/schedule of their latest cycle on protocol A8641014. PF-03084014 will be administered twice a day in the morning and evening divided by approximately 12 hours. PF-03084014 should be administered in cycles of 21 days continuously.
  Other Names: Gamma Secretase Inhibitor

SUMMARY:
This is a single-center, open label, non randomized, compassionate use protocol in patients with advanced solid tumor malignancies who were previously enrolled in the phase I study (NCT00878189) of this agent.

DETAILED DESCRIPTION:
This is an expanded access-physician sponsored trial of PF-03084014, a novel gamma-secretase inhibitor being developed for cancer therapy. This trial is designed for patients who have been on a previous Industry-sponsored phase I trial using PF-03084014 for> 1 year. The study is designed to evaluate the safety of prolonged oral administration of single agent PF-03084014. There are two study subjects with desmoid tumor who have been on the trial for a prolonged period of time (54 and 77 months, respectively) with either stable disease or response, indicating significant clinical benefit for a patient population in which there are few options. The goal of this protocol is to allow these subjects, who are clearly benefiting from PF-03084014, to continue to receive it

ELIGIBILITY:
Inclusion Criteria:

- Patients who are currently enrolled in A8641014 for > 1 year are eligible

Exclusion Criteria:

* Prior treatment with a gamma secretase inhibitor for treatment of cancer
* Patients taking Tamoxifen
* Patients with active graft versus host disease
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
* Patients who are pregnant or breast-feeding
* Patients with clinical evidence of central nervous system disease

Ages: 16 Years to 101 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Wells Messersmith, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States